CLINICAL TRIAL: NCT03800264
Title: Bisoprolol Versus Corticosteroid and Bisoprolol Combination for Prophylaxis Against Atrial Fibrillation After on Pump Coronary Artery Bypass Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Bisoprolol vs corticosteroi
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Prevention; Atrial Fibrillation; CABG
Keywords: Bisoprolol,; corticosteroid,; atrial fibrillation; cardiac surgery
MeSH Terms: conditions — Atrial Fibrillation | interventions — Bisoprolol; Hydrocortisone

STUDY DESIGN:
Intervention Model Description: DOUBLE BLINDED RANDOMIZED STUDY
Who Masked: Participant
Masking Description: BLINDED
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BISOPROLOL (Active Comparator): BISOPROLOL 5mg per oral (P.O.) in the evening of the operation and then one dose (5 mg) every twenty four hours during the next two days.
  Interventions: Drug: Bisoprolol
- hydrocortisone (Active Comparator): hydrocortisone 100 mg intravenously is given in the evening of the operation and then 100 mg every eight hours during the next two days.
  Interventions: Drug: Bisoprolol

INTERVENTIONS:
Drug: Bisoprolol — PREVENTIVE DOUBLE BLINDED
  Other Names: HYDROCORTISONE

SUMMARY:
Background: Atrial fibrillation (AF) is the most common cardiac arrhythmia that occurs after on pump coronary artery bypass graft (CABG) surgery. It is associated with postoperative complications, including increased risk of stroke, prolonged hospital stay and increased costs.

Objectives: The aim of this study was to find reliable, effective, safe and well tolerated tools for the prevention of AF after on pump coronary artery bypass surgery.

Patients and methods: The study included 176 patients (age range 40 to 79 years) and scheduled for elective on pump CABG operations without concomitant procedures. The patients were divided randomly into two equal groups. Group (A) in which bisoprolol was used for prophylaxis against atrial fibrillation after surgery. Group (B) in which bisoprolol and hydrocortisone were used for prophylaxis against atrial fibrillation after surgery. For each patient, the following data were collected: gender, preoperative diseases, intraoperative cross clamp time, cardiopulmonary bypass time, and Lt internal mammary Artery usage, incidence of postoperative atrial fibrillation, death, myocardial infarction chest infection and C - reactive protein levels.

DETAILED DESCRIPTION:
The study was conducted at The Cardiothoracic surgery intensive care unit of Ain Shams University hospitals during a period of 6 months. The study protocol was approved by "research and ethics committee" of anesthesia and intensive care department, Ain Shams University. Informative consent was obtained from the patients before enrolling in the study.

176 Patients were registered in the study. Patients were randomly allocated by computer-generated random number list into two study groups of 88 patients each, with a range of age between 40 and 79 years old and were undergoing elective on pump CABG operations without concomitant procedures.

Group A:

Patients received bisoprolol 5mg per oral (P.O.) in the evening of the operation and then one dose (5 mg) every twenty four hours during the next two days.

Group B:

Patients received bisoprolol as group (A) in addition hydrocortisone 100 mg intravenously is given in the evening of the operation and then 100 mg every eight hours during the next two days.

Exclusion criteria for the study included: Patients with preoperative rhythm abnormalities (sick sinus syndrome, atrioventricular conduction abnormalities, history of chronic or intermittent AF), pretreatment with classes I and III antiarrhythmic agents, receiving anti-hypertensive drugs except angiotensin convertor enzyme (ACE) inhibitors, thyroid disease, renal or liver disease, peripheral arterial atherosclerotic disease, thrombophlebitis, uncontrolled diabetes mellitus, systemic bacterial or mycotic infection, active tuberculosis, Cushing's syndrome, peptic ulcer, psychotic mental disorder, Herpes Simplex keratitis and chronic obstructive pulmonary disease were not included in the study.

Intraoperative technique:

After sedation with diazepam (10 mg intramuscular), radial arterial catheterization, intravenous catheters, and a central venous catheter were introduced in the operating theater. Hemodynamic parameters; Heart rate monitoring, mean arterial pressure, rectal temperature, central venous pressure and arterial blood gas throughout the process was observed. Anesthesia was started by fentanyl (35 mg / kg) and muscle relaxation was achieved with pancronium (0.1 mg / kg), then endotracheal intubation using ventilation with 100% oxygen. The median incision of the sternum was used for cardiac exposure. The left internal mammary artery was harvested and the saphenous vein was prepared, if necessary. All operations were performed under cardiopulmonary bypass and moderate hypothermia (28-328C) with flow rates of 2.2-2.4 l / m2 and the mean perfusion pressure of 50-85 mm Hg. Heart failure was assisted by initial crystalloid cardioplegia (48C, 15 cc / kg) and heart preservation was assisted with 400 cc cold blood Cardioplegia every 20 minutes. The hot shut was performed shortly before removing the cross clamp. The venous cannula was inserted through the right atrial appendix. The arterial cannula was placed in the ascending aorta.

2.3. Postoperative Monitoring: All patients were continuously monitored at the ICU with electrocardiography (ECG), invasive blood pressure and with finger probe for oxygen saturation within 48 h.

Patients developed atrial fibrillation received treatment according to their condition, if they are haemodynamically unstable electrical cardioversion (synchronized adjusted at 100 joules using biphasic electrical cardiovertor) was applied. If they are haemodynamically stable pharmacological cardioversion (amiodarone 5 mg/kg intravenous over 60 minutes, then 1.2 grams per day by continuous intravenous infusion) was used. (5)

ELIGIBILITY:
Inclusion Criteria:

- .176 Patients were registered in the study.

.Range of age between 40 and 79 years old .Undergoing elective on pump CABG operations without concomitant procedures.

Exclusion Criteria:

* : Patients with preoperative rhythm abnormalities (sick sinus syndrome,

  * atrioventricular conduction abnormalities,
  * history of chronic or intermittent AF),
  * pretreatment with classes I and III antiarrhythmic agents,
  * receiving anti-hypertensive drugs except angiotensin convertor enzyme (ACE) inhibitors,
  * thyroid disease,
  * renal or liver disease,
  * peripheral arterial atherosclerotic disease,
  * thrombophlebitis,
  * uncontrolled diabetes mellitus,
  * systemic bacterial or mycotic infection,
  * active tuberculosis,
  * Cushing's syndrome,
  * peptic ulcer,
  * psychotic mental disorder,
  * Herpes Simplex keratitis
  * chronic obstructive pulmonary disease were not included in the study.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
HEART RATE | two days
  atrial fibrillation

CONTACTS AND LOCATIONS:
Locations (1):
- Ramymahrose, Cairo, Egypt